CLINICAL TRIAL: NCT06652412
Title: Comprehensive Geriatric Assessment (CGA) Guided Ultrafractionated Radiotherapy and Systemic Treatment in Elderly or Frail Patients with Inoperable Localized Colorectal Cancer
Brief Title: CGA Guided Ultrafractionated RT and Systemic Treatment in Elderly or Frail Patients with Inoperable Localized CRC
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Zhen Zhang, Principal Investigator, Fudan University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FDRT-2024-137-3690
Record Dates: First submitted 2024-10-21; First posted 2024-10-22 (Actual); Last update posted 2024-10-28 (Actual); Status verified 2024-10

CONDITIONS: Colon Cancer; Rectal Cancer
MeSH Terms: conditions — Colonic Neoplasms; Rectal Neoplasms | interventions — sintilimab; Fluorouracil; raltitrexed; Oxaliplatin; Irinotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- CGA cohort (Experimental): in cohort 1, all patients will receive Ultrafractionated RT, PD-1 antibody, and Comprehensive Geriatric Assessment (CGA) Guided systemic treatment.
  Furthermore, CGA will assess all patients and classify them into Frail, Vulnerabe, or Fit. Frail patients will receive Best Supportive Care (BSC); Vulnerabe patients will receive single agent chemotherapy and BSC; Fit patients will receive doublet chemotherapy and BSC.
  Interventions: Drug: Ultrafractionated RT and CGA Guided systemic treatment.; Radiation: Ultrafractionated Radiotherapy; Drug: Sintilimab; Drug: Fluorouracil; Drug: Raltitrexed; Drug: Oxaliplatin; Drug: Irinotecan (CPT-11)
- external control cohort (Other): external control from real word, data of patients with the same baseline characteristics from the same period and the same institute will be prospectively collected.
  Interventions: Other: data prospectively collected

INTERVENTIONS:
Drug: Ultrafractionated RT and CGA Guided systemic treatment. — in cohort 1, all patients will receive Ultrafractionated RT (1Fx every 3 or 4weeks) and Sintilimab (q3w). Furthermore, CGA will assess all patients and classify them into Frail, Vulnerabe, or Fit. Frail patients will receive Best Supportive Care (BSC); Vulnerabe patients will receive Fluorouracil/Raltitrexed and BSC; Fit patients will receive Fluorouracil/Raltitrexed, Oxaliplatin/Irinotecan, and BSC.
  Arms: CGA cohort
Other: data prospectively collected — in cohort 2, external control from real word, data of patients with the same baseline characteristics from the same period and the same institute will be prospectively collected.
  Arms: external control cohort
Radiation: Ultrafractionated Radiotherapy — 1Fx every 3 or 4weeks
  Arms: CGA cohort
Drug: Sintilimab — 200 mg q3w
  Arms: CGA cohort
Drug: Fluorouracil — 5-Fluorouracil or capecitabine
  Arms: CGA cohort
Drug: Raltitrexed — Raltitrexed
  Arms: CGA cohort
Drug: Oxaliplatin — Oxaliplatin
  Arms: CGA cohort
Drug: Irinotecan (CPT-11) — irinotecan
  Arms: CGA cohort

SUMMARY:
This is a prospective, multicentre, cohort study. For cohort 1, experimental cohort, older or Frail patients with inoperable localized colorectal cancer will receive Ultrafractionated Radiotherapy (RT) and Comprehensive Geriatric Assessment (CGA) Guided systemic treatment. All patients will receive Ultrafractionated RT and PD-1 antibody. Furthermore, CGA will assess all patients and classify them into Frail, Vulnerabe, or Fit. Frail patients will receive Best Supportive Care (BSC); Vulnerabe patients will receive Fluorouracil/Raltitrexed and BSC; Fit patients will receive Fluorouracil/Raltitrexed, Oxaliplatin/Irinotecan, and BSC.

For cohort 2, external control from real word, data of patients with the same baseline characteristics from the same period and the same institute will be prospectively collected.

The primary endpoint is complete response (CR, pathological complete response [pCR] plus clinical complete response [cCR]) rate. The secondary endpoints include the grade 3-4 acute adverse effects rate, anal preservation rate, survival etc.

DETAILED DESCRIPTION:
This is a prospective, multicentre, cohort study. For cohort 1, experimental cohort, older or Frail patients with inoperable localized colorectal cancer will receive Ultrafractionated Radiotherapy (RT) and Comprehensive Geriatric Assessment (CGA) Guided systemic treatment. All patients will receive Ultrafractionated RT and PD-1 antibody. Furthermore, CGA will assess all patients and classify them into Frail, Vulnerabe, or Fit. Frail patients will receive Best Supportive Care (BSC); Vulnerabe patients will receive Fluorouracil/Raltitrexed and BSC; Fit patients will receive Fluorouracil/Raltitrexed, Oxaliplatin/Irinotecan, and BSC.

For cohort 2, external control from real word, data of patients with the same baseline characteristics from the same period and the same institute will be prospectively collected.

The primary endpoint is complete response (CR, pathological complete response [pCR] plus clinical complete response [cCR]) rate. The secondary endpoints include the grade 3-4 acute adverse effects rate, anal preservation rate, 1-year DFS rate, 1-year DSS rate, 1-year OS rate etc.

ELIGIBILITY:
Inclusion Criteria:

1. ≥70y, or, ≥60 and <70y but ECOG≥2;
2. male or female;
3. Pathologically confirmed Colorectal adenocarcinoma;
4. any distance from anal verge;
5. Clinical stage ≥T2 and/or N+, without distance metastases;
6. refuse radical operation, physiologically or technically inoperable;
7. No previous radiotherapy in the same field；
8. No chemotherapy prior to enrollment;
9. No immunotherapy prior to enrollment;
10. With good compliance during the study
11. Signed written informed consent

Exclusion Criteria:

1. Known history of other malignancies within 3 years，except cured skin cancer, cervical cancer in situ or thyroid carcinoma.
2. Individuals with a history of uncontrolled epilepsy, central nervous system disease, or psychiatric disorders that, in the judgment of the investigator, are of such clinical severity that they may prevent the signing of an informed consent form or affect the patient's adherence to oral medications
3. Individuals with clinically serious (i.e., active) heart disease, such as symptomatic coronary artery disease, New York Heart Association (NYHA) class II or worse congestive heart failure or severe arrhythmia requiring pharmacologic intervention, or history of myocardial infarction within the last 12 months
4. Individuals with a history of organ transplantation requiring immunosuppressive therapy and long-term hormone therapy
5. Individuals with autoimmune diseases
6. Individuals with severe uncontrolled recurrent infections, or other severe uncontrolled concomitant diseases
7. Baseline hematology and biochemistry did not meet the following criteria: Hb≥90g/L; NEU ≥1.5×109/L; PLT ≥100×109/L; ALT, AST ≤2.5 times the upper limit of normal; ALP ≤2.5 times the upper limit of normal; TB <1.5 times the upper limit of normal; Cr <1 time the upper limit of normal; Alb ≥30g/L
8. Individuals allergic to any drug component of the study

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Estimated)
Dates: Start 2024-11 (Estimated); Primary Completion 2027-11 (Estimated); Study Completion 2028-11 (Estimated)

PRIMARY OUTCOMES:
Complete response (CR) rate | 1 month after the surgery or the decision of W&W
  Rate of complete response (CR), including the rate of pathologic complete response (pCR) after surgery and the rate of clinical complete response (cCR) with Watch & Wait (W&W) strategy.

SECONDARY OUTCOMES:
Grade 3-4 adverse effects rate | From date of randomization until 3 months after the completion neoadjuvant therapy
  Rate of chemotherapy, radiotherapy and immunotherapy related adverse events
1 year anal preservation rate | From date of randomization until the date of or date of death from any cause, whichever came first, assessed up to 12 months.
  1 year anal preservation rate
health-related quality of life (HRQOL) | baseline, and at 3, 6 and 12 months.
  HRQOL assessed with validated European Organisation for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire (QLQ) ColoRectal cancer (CR) with 29 items (C29) and with 30 items (C30). Multiple measurements and scores will be aggregated to arrive at one reported value. Scores at different time points after randomization will be compared to baseline scores.
1 year disease free survival rate | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 12 months.
  Rate of 1 year disease free survival
1 year local recurrence free survival rate | From date of randomization until the date of first documented pelvic failure, assessed up to 12 months.
  Rate of 1 year local recurrence free survival
1 year Disease-specific survival rate | From date of randomization until the date of death from the specific disease, assessed up to 12 months.
  rate of 1 year Disease-specific survival
1 year overall survival rate | From date of randomization until the date of death from any cause, assessed up to 12 months.
  Rate of 1 year overall survival

CONTACTS AND LOCATIONS:
Overall Officials: Zhen ZHANG Principal Investigator, Principal Investigator — Fudan University